CLINICAL TRIAL: NCT05988086
Title: Evaluation of Using Platelet Rich Fibrin Versus Collagen Membrane for Enhancing Healing of Secondary Grafted Alveolar Cleft
Brief Title: Double Closure of Nasal Layer in Alveolar Cleft Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Marwa Taha Ibrahim, lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-OS-9-22-1
Record Dates: First submitted 2023-07-20; First posted 2023-08-14 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Alveolar Cleft
Keywords: alveolar cleft; collagen membrane; platelet rich fibrin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: platelet rich fibrin (Active Comparator): Group 1: This will include 12 children in whom nasal layer of alveolar cleft will be repaired using autologous platelet rich fibrin with autogenous chin bone.
  Interventions: Procedure: platelet rich fibrin
- Group 2:collagen membrane (Active Comparator): Group 2: This will include 12 children in whom nasal layer of alveolar cleft will be repaired using collagen membrane with autogenous chin bone.
  Interventions: Procedure: collagen membrane

INTERVENTIONS:
Procedure: platelet rich fibrin — 12 children in whom nasal layer of alveolar cleft will be repaired using autologous platelet rich fibrin with autogenous chin bone.
  Arms: Group 1: platelet rich fibrin
Procedure: collagen membrane — 12 children in whom nasal layer of alveolar cleft will be repaired using collagen membrane with autogenous chin bone.
  Arms: Group 2:collagen membrane

SUMMARY:
The aim of this prospective study is to evaluate both clinically and radiologically the efficacy of using autologous platelets rich fibrin versus collagen membrane for nasal layer closure in secondary alveolar cleft repair.

DETAILED DESCRIPTION:
Patients and methods: Twenty-four patients with alveolar clefts will be included in this study. The patients will be evaluated with age ranging between (7 - 12) years. The patients will be received, clinically and radiologically examined, and managed at the Oral and Maxillofacial surgery Department, Faculty of Dentistry, Tanta University.

The selected children should possess the following criteria: Their permanent canines either not or partially erupted, has no systemic disorder which can affect the grafting outcome and healing process such as juvenile diabetes mellitus, kidney, liver, or blood diseases and has no associated craniofacial syndromes. The patients will be classified into two groups according to incorporation of autologous platelet rich fibrin or collagen membrane for nasal layer closure with the grafting material, as follow: Group 1: This will include 12 children in whom nasal layer of alveolar cleft will be repaired using autologous platelet rich fibrin with autogenous chin bone. Group 2: This will include 12 children in whom nasal layer of alveolar cleft will be repaired using collagen membrane with autogenous chin bone.

Preoperative evaluation of alveolar cleft site:

all patients will be examined clinically and radiologically. Clinical examination: This will consider the stability of maxillary segments, presence of old scar, asymmetry of the alar base, presence of oronasal fistula, and the presence of erupting teeth in the cleft.

Radiological examination: Panoramic radiographs will be done for each patient and examined as regard: the morphology of the cleft area, the size of the cleft side, the presence or absence of permanent lateral incisor and canine, the development of root length, and stage of eruption of permanent canine and lateral incisor. In addition, Axial computed tomography (CT) scans will be done for each patient to assess and measure local bone mineral density of grafted alveolar bone cleft.

Postoperative evaluation of the grafted site:

The grafted site will be evaluated clinically for healing condition at the follow up periods (1st week, then 1st , 3rd ,6th ,and 9th month postoperatively) ; regarding the presence of inflammation or infection , the soft tissue scar overlying the bone graft , tenderness of bone graft site , recurrence of oronasal fistula , alveolar ridge contour in cleft region and eruption of cleft related teeth . Radiological evaluation will be done for each patient using Axial computed tomography (CT) scans at the follow up period (3rd and 9th month postoperatively) to assess and measure local bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

1. patients with unilateral alveolar cleft
2. the patient's permenant canines either not or partially erupted
3. medically free patients

Exclusion Criteria:

1. patients with bilateral alveolar cleft
2. medically compromised patients
3. Any associated craniofacial syndromes.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | 1 month
  0 representing no pain and 10 representing the highest level of pain
inflammation score scale | 1 month
  0 no inflammation, 1-3 mild inflammation,4-7 moderate inflammation,8-10 severe inflammation
density of bone | 1 month
  density of bone to measure (D1,D2,D3,D4) Frome 150HU to 1250HU

SECONDARY OUTCOMES:
bone mineral density. | 9 months
  density of bone to measure (D1,D2,D3,D4) Frome 150HU to 1250HU

CONTACTS AND LOCATIONS:
Overall Officials: Marwa T Ibrahim, lecturer, Principal Investigator — Tanta University
Locations (1):
- Egypt, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No